CLINICAL TRIAL: NCT01466010
Title: Treatment Outcome After Surgical Treatment of Osteoid Osteoma, a Retrospective Study
Brief Title: Treatment Outcome After Surgical Treatment of Osteoid Osteoma
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S53583
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-09

CONDITIONS: Osteoid Osteoma
Keywords: osteoma, osteoid; surgical procedures, operative; bone neoplasms
MeSH Terms: conditions — Osteoma, Osteoid; Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- osteoid osteoma: patients with osteoid osteoma at any location
  Interventions: Procedure: surgical removal of osteoid osteoma

INTERVENTIONS:
Procedure: surgical removal of osteoid osteoma — surgery for osteoid osteoma: this may include curettage or en-bloc resection of the lesion

SUMMARY:
Purpose of the study:

To retrospectively determine the clinical results in an unselected group of consecutive patients with osteoid osteoma treated by surgery.

Materials and Methods:

In 150 consecutive patients with clinical and/or radiological evidence for osteoid osteoma at any location, the clinical symptoms and imaging findings (radiographs and computed tomography (CT)) were assessed before and after surgery. There were no exclusion criteria for this study. A good response was defined as disappearance of symptoms that were manifested at presentation and were attributed to osteoid osteoma. Clinical assessment after the procedure was performed prior to discharge; within 2 weeks after the procedure; and at 3, 6, and 12 months follow-up. After 24 months, a postal questionnaire was used for assessment. Radiographic evaluation (radiographs and thin-slice CT) was performed routinely pre-operatively and one year after surgery.

In case of persisting or recurring symptoms the follow-up protocol was again performed according to the initial protocol.

All patients gave their informed consent both for the surgical intervention as for the use of their patient data in this retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* patient with osteoid osteoma at any location.

Exclusion Criteria:

* none.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with osteoid osteoma at any location.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 1998-01; Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven Dept of Radiology, Leuven, Vlaams Brabant, Belgium